CLINICAL TRIAL: NCT06217536
Title: Phase 1b/2 Trial Using Neoadjuvant Lurbinectedin With Concurrent Preoperative Radiation in Patients With Locally Advanced Soft Tissue Sarcomas of Extremity, Trunk, and Retroperitoneum
Brief Title: Neoadjuvant Lurbinectedin and Preoperative Radiation for Treating Soft Tissue Sarcomas
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: University of California, San Francisco (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23872; NCI-2024-00107 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Locally Advanced Soft Tissue Sarcoma
MeSH Terms: interventions — PM 01183; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1b, Cohort 1 (Extremity and Trunk Sarcoma) (Experimental): Participants will receive up to 3.2 mg/m^2 of neoadjuvant lurbinectedin IV once every cycle (a cycle is 21 days) in combination with 2 weeks of pre-operative radiation given as 35 Gy in 5 fractions (gross tumor volume (GTV)) with fractions administered at least every other day starting on cycle 2 for participants with extremity and trunk sarcoma. Non-investigational surgery will take place 4-6 weeks after completion of radiation therapy. Participants with metastatic disease at the time of study enrollment may be able to continue study treatment for 2 years from the time of initiating treatment. Participants with localized disease at the time of study enrollment may continue study treatment for approximately 3 months AND then be followed on-study surveillance.
  Interventions: Drug: Lurbinectedin; Radiation: Radiotherapy; Procedure: Non-investigational surgery
- Phase 1b, Cohort 2 (Extremity Myxoid Liposarcoma) (Experimental): Participants will receive up to 3.2 mg/m^2 of neoadjuvant lurbinectedin IV once every cycle (a cycle is 21 days) in combination with 2 weeks of pre-operative radiation given as 35 Gy in 5 fractions (gross tumor volume (GTV)) with fractions administered at least every other day starting on cycle 2 for participants with extremity myxoid Liposarcoma. Non-investigational surgery will take place 4-6 weeks after completion of radiation therapy. Participants with metastatic disease at the time of study enrollment may be able to continue study treatment for 2 years from the time of initiating treatment. Participants with localized disease at the time of study enrollment may continue study treatment for approximately 3 months AND then be followed on-study surveillance.
  Interventions: Drug: Lurbinectedin; Radiation: Radiotherapy; Procedure: Non-investigational surgery
- Phase 1b, Cohort 3: Retroperitoneal Sarcoma (Experimental): Participants will receive up to 3.2 mg/m^2 of neoadjuvant lurbinectedin IV once every cycle (a cycle is 21 days) in combination with 6 weeks of pre-operative conventional external beam radiation therapy given as 45-50.4 Gy delivered over 25-28 fractions starting on cycle 1 for participants with retroperitoneal sarcoma. Non-investigational surgery will take place 4-6 weeks after completion of radiation therapy. Participants with metastatic disease at the time of study enrollment may be able to continue study treatment for 2 years from the time of initiating treatment. Participants with localized disease at the time of study enrollment may continue study treatment for approximately 3 months AND then be followed on-study surveillance.
  Interventions: Drug: Lurbinectedin; Radiation: Radiotherapy; Procedure: Non-investigational surgery
- Phase 2, Cohort 1: Extremity and trunk sarcoma (Experimental): Participants will receive the maximum tolerated dose of neoadjuvant lurbinectedin IV once every cycle (a cycle is 21 days) in combination with 2 weeks of pre-operative radiation given as 35 Gy in 5 fractions (gross tumor volume (GTV)) with fractions administered at least every other day starting on cycle 2 for participants with extremity and trunk sarcoma. Non-investigational surgery will take place 4-6 weeks after completion of radiation therapy. Participants with metastatic disease at the time of study enrollment may be able to continue study treatment for 2 years from the time of initiating treatment. Participants with localized disease at the time of study enrollment may continue study treatment for approximately 3 months AND then be followed on-study surveillance.
  Interventions: Drug: Lurbinectedin; Radiation: Radiotherapy; Procedure: Non-investigational surgery
- Phase 2, Cohort 2: Extremity myxoid liposarcoma (Experimental): Participants will receive the maximum tolerated dose of neoadjuvant lurbinectedin IV once every cycle (a cycle is 21 days) in combination with 2 weeks of pre-operative radiation given as 35 Gy in 5 fractions (gross tumor volume (GTV)) with fractions administered at least every other day starting on cycle 2 for participants with extremity myxoid Liposarcoma. Non-investigational surgery will take place 4-6 weeks after completion of radiation therapy. Participants with metastatic disease at the time of study enrollment may be able to continue study treatment for 2 years from the time of initiating treatment. Participants with localized disease at the time of study enrollment may continue study treatment for approximately 3 months AND then be followed on-study surveillance.
  Interventions: Drug: Lurbinectedin; Radiation: Radiotherapy; Procedure: Non-investigational surgery
- Phase 2, Cohort 3: Retroperitoneal sarcoma (Experimental): Participants will receive the maximum tolerated dose of neoadjuvant lurbinectedin IV once every cycle (a cycle is 21 days) in combination with 6 weeks of pre-operative conventional external beam radiation therapy given as 45-50.4 Gy delivered over 25-28 fractions starting on cycle 1 for participants with retroperitoneal sarcoma. Non-investigational surgery will take place 4-6 weeks after completion of radiation therapy. Participants with metastatic disease at the time of study enrollment may be able to continue study treatment for 2 years from the time of initiating treatment. Participants with localized disease at the time of study enrollment may continue study treatment for approximately 3 months AND then be followed on-study surveillance.
  Interventions: Drug: Lurbinectedin; Radiation: Radiotherapy; Procedure: Non-investigational surgery

INTERVENTIONS:
Drug: Lurbinectedin — Given intravenously (IV)
  Other Names: Zepzelca
Radiation: Radiotherapy — Conventionally fractionated radiotherapy or external beam radiation
  Other Names: Radiation therapy
Procedure: Non-investigational surgery — Non-investigational surgical procedure on tumor tissue

SUMMARY:
This is a multi-center, multi-arm open-label phase Ib/II clinical study assessing the efficacy of concurrent lurbinectedin in combination with radiotherapy in patients with locally advanced, resectable, high-grade sarcomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Phase Ib:

I. To determine the safety and tolerability of neoadjuvant lurbinectedin

* in combination with preoperative 2 weeks of hypofractionated radiation for extremity and trunk sarcoma, or
* with 6 weeks of conventionally fractionated radiation for retroperitoneal sarcoma II. To determine the maximum tolerated dose (MTD) for neoadjuvant lurbinectedin in combination with preoperative external beam radiation therapy (EBRT) in patients with sarcoma.

Phase II:

I. To estimate the efficacy of neoadjuvant lurbinectedin in combination with preoperative EBRT (hypofractionated or conventionally fractionated), according to endpoint defined by sarcoma type and location:

* Cohort 1: extremity and trunk sarcoma (HFRT)
* Cohort 2: Extremity myxoid liposarcoma (HFRT)
* Cohort 3: Retroperitoneal sarcoma (CFRT course)

SECONDARY OBJECTIVES:

I. Time to disease progression (local or distant recurrence).

II. Overall response rate (ORR) pre-operative as measured by RECIST 1.1 or a later tool for monitoring disease progression.

III. Overall survival.

IV. To grade radiation related skin toxicity overlying the tumor area.

V. To determine long term major wound healing complications with the use of this combination in all cohorts.

EXPLORATORY OBJECTIVES:

I. To evaluate changes in monocyte, macrophage, T cell, and RNA expression levels over time.

OUTLINE:

Participants will receive neoadjuvant lurbinectedin concurrent with radiation therapy. Non-investigational surgery will be performed 4-6 weeks from the end of radiation therapy. Participants with localized disease at the time of study enrollment will be on surveillance on-study for 2 years. Post-operatively participants will be followed every 12 +/- 4 weeks for approximately 2 years from the end of treatment. Participants with known metastatic disease will be followed until progression, toxicity and thereafter for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Must have histologically or cytologically confirmed diagnosis of locally advanced soft tissue sarcoma of extremity, trunk or retroperitoneum that is resectable and for which preoperative radiotherapy is considered appropriate.

   1. Including metastatic (stage IV) disease for which radiotherapy and surgical resection of the primary tumor are indicated.
   2. Grade 1 myxoid liposarcoma can be included if preoperative radiotherapy is considered appropriate.
   3. For all other sarcomas, only grade 2 or 3 will be included.
2. Those with locally recurrent sarcoma after surgery alone are eligible for enrollment if other inclusion criteria are met.
3. Must have measurable disease defined as a tumor size at least >= 5 cm in the longest diameter as measured by Computerized tomography (CT) scan or Magnetic resonance imaging (MRI) for which radiation is feasible and indicated.
4. Age >=18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status <= 1 (Karnofsky ≥ 70%).
6. Demonstrates adequate organ function within 21 days of Day 1 as defined below:

   1. Hemoglobin >= 9.0 g / dL.
   2. prothrombin time (PT) (or International Normalized Ratio (INR)) and partial thromboplastin time (PTT) (or activated partial thromboplastin time (aPTT)) <1.5 x upper limit of normal (ULN).
   3. Absolute neutrophil count >=1,500/microliter (mcL).
   4. Platelets >=100,000/mcL.
   5. Total bilirubin within normal institutional limits, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits.
   6. Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT)<=3 X institutional upper limit of normal.
   7. Alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) <=3 X institutional upper limit of normal.
   8. Alkaline phosphatase (ALP) < 2.5 × ULN.
   9. Creatinine <= 2 x within institutional upper limit of normal OR creatinine clearance Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2, calculated using the Cockcroft-Gault equation, unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
9. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
10. Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured. For individuals with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
11. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
12. The effects of Lurbinectedin on the developing human fetus are unknown. For this reason and because Lurbinectedin used in this trial are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (2 methods of contraception including hormonal and barrier method of birth control) for the duration of study participation and for 6 months after last administration of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. A female is considered to be of childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) if she meets the following criteria:

    * is postmenarchal,
    * has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and
    * has not undergone surgical sterilization (removal of ovaries and/or uterus). - Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after last administration of study treatment.

Exclusion Criteria:

1. Has the following histologic subtypes: gastrointestinal stromal tumor (GIST), desmoid, Ewing sarcoma, bone sarcomas, Kaposi sarcoma.
2. Prior history of trabectedin or lurbinectedin treatment.
3. Prior radiation therapy in excess of 20 Gray (Gy) conventionally fractionated radiotherapy (RT) to the site of the current diagnosis of sarcoma. No overlap with prior radiation fields in excess of 20 Gy is allowed.
4. Currently receiving treatment in another invasive investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s).
5. Known central nervous system (CNS) disease, except for treated brain metastasis: Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS); Gamma Knife, linear particle accelerator (LINAC), or equivalent) or a combination as deemed appropriate by the treating physician. Participants with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to lurbinectedin.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Participants on strong or moderate cytochrome P450 (CYP)3A inducers or inhibitors and cannot be substituted for other drugs.
9. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this study.
10. Has received systemic anti-cancer therapies within 3 weeks of first dose, radiation within 2 weeks, or antibody therapy within 4 weeks. Concomitant administration of Luteinizing hormone-releasing hormone (LHRH) analogues for prostate cancer and somatostatin analogues for neuroendocrine tumors are allowed as per standard of care.
11. Has not recovered from adverse events due to prior anti-cancer therapy to <= grade 1 or baseline (other than alopecia).
12. Is currently receiving any other investigational agents.
13. Any concurrent illness in the opinion of the investigator would affect treatment compliance.
14. Participants needing concurrent antiemetic aprepitant or any other Neurokinin 1 (NK1) antagonist or related Substance P-antagonists (except rolapitant).
15. Pregnant participants are excluded from this study because lurbinectedin has the potential for teratogenic or abortifacient effects. Females of childbearing potential (definition as above) must undergo a urine pregnancy test per institutional guidelines within 7 days prior to Day 1 of study treatment. Participants with a positive urine pregnancy test are excluded.
16. Breast-feeding participants are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lurbinectedin, breastfeeding should be discontinued if the mother is treated with lurbinectedin and for 2 weeks after the last dose.
17. Participants of childbearing potential who are unwilling to use at least 2 highly effective methods of contraception during study treatment and for 90 days following the last dose of study treatment.
18. Participants with a known history of collagen vascular disease on active therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with dose-limiting toxicities (DLTs) (Phase 1b) | 4 weeks
  The proportion of participants with reported DLTs will be reported for
Maximum Tolerated Dose (MTD) (Phase 1b) | Up to 6 months
  MTD is defined as the highest dose at which no more than one instance of dose limiting toxicity (DLT) is observed among 1 of 6 participants treated.
Pathological necrosis rate (Phase 2, Cohort 1) | Up to 12 weeks
  Pathological necrosis rate, defined as the proportion of participants with >=95% pathological necrosis.
Local control rate (Phase 2, Cohort 2) | Up to 12 weeks
  Local control rate is defined as the proportion of participants with >=50% of the resected sample showing any histological treatment effect.
Overall response rate (Phase 2, Cohort 3) | Up to 12 weeks
  Overall response rate is defined as the proportion of participants with a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Median time to disease progression (TTP) | Up to 2 years
  Time to progression is defined as the time from first day of study treatment to first documented occurrence of disease progression (including local and distant recurrences). Participants without progression will be censored at their last disease evaluation will be reported.
Overall Response Rate (ORR) | Up to 12 weeks
  The proportion of pre-operative participants with a confirmed CR or PR as measured by RECIST 1.1 or a later tool for monitoring disease progression will be reported.
Median Overall Survival (OS) | Up to 2 years
  The median overall survival time is defined as the time from first day of study treatment to death due to any cause will be reported. Participants who are still alive will be censored at their last date known to be alive.
Incidence of radiation related skin toxicity | Up to 6 months
  Incidence of radiation related skin toxicity by grade as classified by the NCI CTCAE version 5.0 and additionally assessed by radiation oncologists will be reported.
Proportion of participants requiring wound care | Up to 4 months after non-investigational surgery
  The proportion of participants requiring secondary operation under general or regional anesthesia for wound repair, invasive procedure without general or regional anesthesia (mainly aspiration of seroma), readmission for wound care such as intravenous antibiotics, or persistent deep packing for 120 days (4 months) or longer will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Varun Monga, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No